CLINICAL TRIAL: NCT06515678
Title: Impact of Antihypertensive Therapy on Recurrence Risk of Ovarian Cancer for Patients Treated With Bevacizumab Maintenance: A Target Trial Emulation
Brief Title: Impact of Antihypertensive Therapy on Recurrence Risk of Ovarian Cancer for Bevacizumab-associated Hypertension
Acronym: IATRO
Status: Active, not recruiting | Type: Observational
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Collaborators: Dr Floriane Jochum, Principal Investigator (Unknown); Institut Curie (Other)
Responsible Party: Principal Investigator, Paul Gougis, Principal Investigator, Groupe Hospitalier Pitie-Salpetriere
Other Study IDs: CIC1421-24-09
Record Dates: First submitted 2024-07-04; First posted 2024-07-23 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Ovarian Cancer; Antiangiogenic-Associated Hypertension; Adjuvant Bevacizumab; Hypertension
Keywords: antiangiogenics; antihypertensive; ovarian cancer surgery; bevacizumab; calcium channel blockers; angiotensin-converting enzyme inhibitors
MeSH Terms: conditions — Ovarian Neoplasms; Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Main analysis - antihypertensive therapy with bevacizumab (ACEi or CCBs): Adjuvant/maintenance bevacizumab after ovarian cancer debulking surgery with antihypertensive therapy monotherapy.
  Any patients with bevacizumab treated with monotherapy ACEi (arm A) or CCB (arm B) up to 6 months following debulking surgery
  Interventions: Drug: arm A - angiotensin converting enzyme inhibitors (ACEi); Drug: arm B - calcium channel blockers (CCBs)
- Complementary group - arm C1 - bevacizumab without antihypertensive therapy: Patients treated with bevacizumab without initiation of antihypertensive treatment within 6 months following debulking surgery
- Complementary group - arm C2 - standard chemotherapy alone: Patients who were only treated by standard chemotherapy within 6 months following debulking surgery without bevacizumab
- Complementarity analysis - 1st-line CCB vs ACEi vs ARBs: Adjuvant/maintenance bevacizumab after ovarian cancer debulking surgery with antihypertensive therapy monotherapy.
  Any patients with bevacizumab treated with Renin Angiotensin Aldosterone System (RAAS) inhibitor drug among ACEi (arm A) versus angiotensin receptor blocker ARB (arm R) versus CCB (arm B)
  Interventions: Drug: arm A - angiotensin converting enzyme inhibitors (ACEi); Drug: arm B - calcium channel blockers (CCBs); Drug: arm R - angiotensin receptor blockers ARB
- Sensitivity analysis: Sensitivity analysis S1 - Impact of Antihypertensive Treatment Switching. The investigators will utilize time-varying inverse probability of censoring weights (IPCW). The first step of the IPCW method consists in censoring patients who interrupt their initially assigned treatment. The second step of the IPCW method is thus to use IPCW with baseline covariates and time-dependent covariates linked to the treatment switching. (i) Number of cardiology consultations, (ii) Number of nephrology consultations or proteinuria, (iii) Number of cardiovascular events related to hypertension (MACE broad)
  Sensitivity analysis S2 - Exclusion of patients with isolated proteinuria or elevated proteinuria: The investigators will reproduce the main analysis, excluding patients with signs of isolated proteinuria or elevated proteinuria.
  Interventions: Drug: arm A - angiotensin converting enzyme inhibitors (ACEi); Drug: arm B - calcium channel blockers (CCBs)

INTERVENTIONS:
Drug: arm A - angiotensin converting enzyme inhibitors (ACEi) — Patients with ACEi monotherapy before or within 6 months following debulking surgery.
  ACEi will be defined as any drugs from the Anatomical Therapeutic Classification C09AA with an indication for hypertension, including but not limited to: captopril, enalapril, lisinopril, perindopril, ramipril, quinapril
  Groups: Complementarity analysis - 1st-line CCB vs ACEi vs ARBs; Main analysis - antihypertensive therapy with bevacizumab (ACEi or CCBs); Sensitivity analysis
Drug: arm B - calcium channel blockers (CCBs) — Patients with CCB monotherapy before or within 6 months following debulking surgery.
  CCBs will be defined as any drugs from the Anatomical Therapeutic Classification C08CA with an indication for hypertension, including but not limited to: amlodipine, felodipine, isradipine, nicardipine, nifedipine
  Groups: Complementarity analysis - 1st-line CCB vs ACEi vs ARBs; Main analysis - antihypertensive therapy with bevacizumab (ACEi or CCBs); Sensitivity analysis
Drug: arm R - angiotensin receptor blockers ARB — Patients with angiotensin receptor blocker (ARB) before or within 6 months following debulking surgery.
  ARBs will be defined as any drugs from the Anatomical Therapeutic Classification C09CA with an indication for hypertension, including but not limited to: losartan, valsartan, irbesartan, candesartan or olmesartan medoxomil.
  Groups: Complementarity analysis - 1st-line CCB vs ACEi vs ARBs

SUMMARY:
Antiangiogenic therapies like bevacizumab, have notably improved cancer treatment, including for gynecological cancers, by inhibiting the vascular endothelial growth factor and thus limiting tumor growth. In treating advanced ovarian cancer, bevacizumab has been shown to extend progression-free survival by four months, though it also induces or worsens hypertension in 2 to 19% of patients by affecting vascular nitric oxide production or by capillary rarefaction. This hypertension may result in severe cardiovascular events, necessitating the use of antihypertensive drugs like calcium channel blockers and RAAS inhibitors (angiotensin converting enzyme - ACE - inhibitors mainly), despite some concerns about their effects on VEGF secretion and CA125 levels. Clinical guidelines vary, with some favoring ACE inhibitors while others recommend calcium channel blockers, underlining the need for comparative studies on these drugs' oncological and cardiovascular impacts. To address these issues, this study utilizes an emulated trial approach, leveraging comprehensive data from the French National Health Data System to compare the efficacy of these antihypertensive classes in reducing relapse and improving survival in ovarian cancer patients treated with bevacizumab.

The investigators will emulate a target clinical trial to compare the impact of antihypertensive treatments on outcomes of patients with bevacizumab-associated hypertension by ACE inhibitors (arm A) versus calcium channel blockers (CCBs, arm B) on the risk of ovarian cancer withdrawal after surgery.

DETAILED DESCRIPTION:
Antiangiogenic therapies, such as bevacizumab, have significantly improved the treatment landscape of various cancers, including gynecological types. Bevacizumab is a humanized monoclonal IgG1 antibody targeting all forms of human vascular endothelial growth factor-A (VEGF), essential for angiogenesis in healthy and cancerous tissues. This drug inhibits angiogenesis primarily by blocking VEGF from activating its receptors, VEGFR, on endothelial cells, thus limiting tumor growth by cutting off their blood supply and aiding the effectiveness of cytotoxic drugs by reducing tumor interstitial pressure and abnormal blood vessels.

For advanced ovarian cancer, bevacizumab was found to improve the median progression-free survival of 4 months. However, targeting tumor vessels will eventually modify the patients' vasculature, leading to hypertension in 2 to 19% of patients as per a meta-analysis. VEGF-VEGFR pathway inhibition can cause hypertension by inhibiting the production of nitric oxide in the arterial wall or by capillary rarefaction and increased afterload. Several retrospective studies support a correlation between the occurrence of a bevacizumab-associated hypertension (BIH) and outcomes, highlighting the link between tumor and patient vasculature. However, bevacizumab-associated hypertension can lead, in some rare cases, to major adverse cardiovascular events (MACE).

Multiple treatments have been proposed to control this adverse reaction. Calcium channel blockers (CCBs) such as amlodipine have been proposed and offers a way to control bevacizumab-associated hypertension. Angiotensin-converting enzyme inhibitors (ACEi), which targets the renin-angiotensin-aldosterone system (RAAS) to control hypertension, could also constitute an interesting option and could be more efficient.

However, there is both caution against the use of CCBs and ACEis, since nifedipine has been shown to induce VEGF secretion in vitro, and ACEi (enalapril and perindopril) have been associated in a case report with CA125 increase.

Current guidelines vary on the preferred class of medication for initial management of antiangiogenic-associated hypertension. The European Society of Cardiology (ESC) guidelines favor ACEis as the first-line treatment, whereas guidelines for gynecological cancers suggest CCBs for managing BIH in patients without other comorbidities. This discrepancy highlights the need for direct comparisons of oncologic and cardiologic outcomes in this context.

Randomized controlled trials (RCTs), despite being the gold standard, face practical and financial constraints that may limit their use. In the absence of RCT, observational data can serve as a crucial alternative for estimating real-world causal effects. However, observational studies come with challenges, such as confounding factors due to the lack of randomization and the risk of immortal-time bias. A recent advancement in addressing these challenges is the use of emulated trials, which strive to replicate the conditions of a target RCT. This approach, employing propensity-score adjustment methods, has shown promise in extracting the highest level of evidence from observational data. The SNDS, covering 98.8% of the French population, offers extensive and detailed demographic, health condition, and healthcare utilization data, enabling a thorough and representative analysis of healthcare outcomes in oncology.

In this study, to address measured confounding at baseline, an exact copy of each patient's record will be created and allocated to each arm of the study, ensuring identical baseline characteristics across the study groups. Clones will be artificially censored when their observed trajectories deviated from the treatment strategy of the arm to which they were assigned. This informative artificial censoring introduces selection bias over time, which will be addressed using inverse probability of censoring (IPC) weights. Standardized mean differences (SMDs) will be derived to assess adjustment quality after IPC weighting.

The per-protocol average treatment effect (ATE) will be estimated by the one- and three-year differences in PFS probability and three-year restricted mean survival time (RMST) differences in the IPC-weighted population. This will be visually assessed using weighted Kaplan-Meier survival curves. Similar steps will be performed for overall survival (OS) at one, three, and five years for survival probability differences, and at five years for RMST.

This study focuses on comparing the effects of antihypertensive drugs - ACEi vs CCBs- on the risk of relapse in patients undergoing adjuvant maintenance treatment with bevacizumab for ovarian cancer after debulking surgery. It employs an emulation of a clinical trial using data from the French National Health Data System (SNDS). Secondary objectives will include examining the causal impact of these antihypertensive classes on overall survival, the incidence of MACE and the time to treatment failure.

ELIGIBILITY:
Inclusion Criteria:

* women with newly ovarian cancer diagnosis (FIGO III to IV)
* age over 18 years old at time of ovarian cancer diagnosis
* diagnosed between January 1, 2011 and December 31, 2020
* with debulking ovarian cancer surgery and adjuvant chemotherapy

Exclusion Criteria:

* not in the "Regime general" "Sécurité Sociale" reimbursement system
* without standard chemotherapy protocol (carbotaxol every 3 weeks or weekly)
* history of heart failure or heart surgery, cardiovascular infarction or any coronaropathy disease, cerebro-vascular disease, arteriopathy of the lower limb, within the year before ovarian cancer surgery. Patients with history of hypertension without any complications were not excluded.
* bevacizumab initiation prior to debulking surgery
* combination of antihypertensive classes prior bevaizumab or as the first-line hypertensive therapy of bevacizumab-associated hypertension
* antihypertensive monotherapy from other classes than CCBs and ACEi (ARBs, beta-blockers, diuretics etc...) as the anti-hypertensive therapy. Therapy could be initiated before ovarian surgery.

Complementary analysis :

- patients treated by ARBs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of women over 18 diagnosed with ovarian cancer between January 1, 2011, and December 31, 2020, who undergone debulking surgery for ovarian cancer with adjuvant chemotherapy.
  In the main target emulated trial, all patients received an antihypertensive first-line monotherapy with either CCBs or ACEi as a stable treatment monotherapy treatment of hypertension prior to bevacizumab or for a bevacizumab-associated hypertension.
  2 complementary cohorts are kept for interpretation and quality control purposes.
Sampling Method: Probability Sample
Enrollment: 9464 (Actual)
Dates: Start 2024-05-20 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival for ovarian cancer | PFS is defined as the time, from ovarian cancer first surgery to death, progression or recurrence, whichever occurres first, assessed up to 7 years
  The per-protocol average treatment effect (ATE) will be estimated by the one-, two-, and three-year differences in PFS probability, and three-year restricted mean survival time (RMST) differences in the IPC-weighted population.
  The main outcome will be at three-year.
  Covariate adjustment :
  Covariates included in the inverse probability weighting are: (i) age at trial inclusion, (ii) number and type of comorbidities, (iii) economic deprivation level, (iv) number of general practitioner consultations the year before, (v) number of gynecologist consultation the year before, (vi) number of cardiology consultation at inclusion, (vii) number of nephrology consultation at inclusion, (viii) FIGO stage, (ix) surgical strategy, (x) hospital annual ovarian cancer volume, and (xi) hospital academic status

SECONDARY OUTCOMES:
Overall survival | OS is defined as the time, from ovarian cancer first surgery to death from any cause, assessed up to 7 years
  The per-protocol average treatment effect (ATE) will be estimated by the one-, two-, three-, and five-year differences in OS probability, and five-year restricted mean survival time (RMST) differences in the IPC-weighted population.
Major Cardiovascular Event (MACE) - narrow definition | Time from ovarian cancer first surgery to the time of MACE-narrow, assessed up to 7 years
  MACE-narrow is defined any acute myocardial infarction or cerebrovascular infarction. A competing risk model will be used for the occurrence of MACE narrow and broad, with death as a competing event. The investigators will utilize time-varying inverse probability of censoring weights (IPCW). The first step of the IPCW method consists in censoring patients who died. The death censoring mechanism may depend on the baseline and time-dependent factors. The IPCW method introduces weights to correct for this dependent censoring. The second step of the IPCW method is thus to use inverse probability of censoring weights with baseline covariates and time-dependent covariates : (i) Number of cardiology consultations, (ii) Number of nephrology consultations. MACE will be analyzed up to 36 months to assess the direct impact of bevacizumab use. Longer-term outcomes will be available in the supplemental only.
Major Cardiovascular Event (MACE) - broad definition | Time from ovarian cancer first surgery to the time of MACE-broad, assessed up to 7 years
  MACE-narrow is defined any acute myocardial infarction or cerebrovascular infarction. A competing risk model will be used for the occurrence of MACE narrow and broad, with death as a competing event. The investigators will utilize time-varying inverse probability of censoring weights (IPCW). The first step of the IPCW method consists in censoring patients who died. The death censoring mechanism may depend on the baseline and time-dependent factors. The IPCW method introduces weights to correct for this dependent censoring. The second step of the IPCW method is thus to use inverse probability of censoring weights with baseline covariates and time-dependent covariates : (i) Number of cardiology consultations, (ii) Number of nephrology consultations. MACE will be analyzed up to 36 months to assess the direct impact of bevacizumab use. Longer-term outcomes will be available in the supplemental only.
Time to treatment failure (TTF) | Time from bevacizumab initiation to the first antihypertensive treatment switch or change to bitherapy, assessed up to 7 years
  Treatment failure is defined as the necessity to switch antihypertensive therapy, add a new antihypertensive therapy (bitherapy), the occurrence of a MACE-broad, recurrence or death. Time to antihypertensive treatment failure (TTF) will be assessed by the median TTF in each study arm (CCBs and ACEi). Dose increase was not considered a treatment failure. TTF is censored at bevacizumab withdrawal.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Institut Curie, Paris
  - Pitié-Salpêtrière, Paris